CLINICAL TRIAL: NCT04950998
Title: A Smartphone Application to Improve Physical Activity in Underactive Older Adults With Mild Cognitive Impairment/Mild Dementia
Brief Title: Smartphone App to Improve Physical Activity in Older Adults With MCI/Mild Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Stacey L. Schepens Niemiec, Associate Professor of Research, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS-19-00444; 3R21AG052838-02S1 (NIH)
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Sedentary Lifestyle; Dementia, Mild; Mild Cognitive Impairment; Memory and Thinking Problems
Keywords: Smartphone app; Physical activity; Older adults
MeSH Terms: conditions — Sedentary Behavior; Dementia; Lymphoma, Follicular; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Target Users - Moving Up-A app (Other): In this single-arm trial, target users (participants) will use a physical activity smartphone app for a two-month period. The app includes motivational messages, tips to increase the intensity level of everyday activities, and strategies to reduce sedentary behaviors. Users can also track their physical activity levels and sedentary activity.
  Interventions: Behavioral: Moving Up - A
- Study Partners - Moving Up-A app (Other): In this single-arm trial, study partners were invited to support target users (participants) in using a physical activity smartphone app for a two-month period. The app includes motivational messages, tips to increase the intensity level of everyday activities, and strategies to reduce sedentary behaviors. Users can also track their physical activity levels and sedentary activity.
  Interventions: Behavioral: Moving Up - A

INTERVENTIONS:
Behavioral: Moving Up - A — Moving Up - A is a physical activity smartphone app for persons with mild cognitive impairment or mild forms of dementia. The app includes a personally tailored set of messages, tips, strategies, and tasks designed to increase physical activity levels and disrupt extended periods of sedentary time. Users also have the ability to track their steps and and sedentary behavior time as well as their progress towards activity goals.

SUMMARY:
The purpose of this study is to develop and test a physical activity-tracking smartphone app designed to facilitate physical activity in older adults with mild cognitive impairments or mild dementia. The app targets provides tips, messages, and strategies to overcome common barriers older adults face to being physically active. Participants will include older adults with memory or thinking problems or those diagnosed with mild cognitive impairment or mild forms of dementia who are smartphone users age 65 years or older and who are not meeting nationally recommended levels of physical activity. In the clinical trial phase of this study, 15 participant-study partner dyads will be oriented to the app and use it for a two-month period. Dyads will keep a diary to document their experiences and participants' activity patterns will also be tracked at the beginning and end of the study. After the two-month app trial is complete, dyads will return for a follow-up interview to discuss their experiences and provide suggestions for app improvements. Findings from this stage of the overall study will be combined with previous study phases to derive specifications for an optimized app for older people with mild cognitive impairments or mild dementia.

ELIGIBILITY:
Inclusion Criteria - Target User:

* 65+ years old
* English speaking;
* resides in local Los Angeles area or the Pacific Time Zone;
* self-reported memory or thinking problems that score within a range of mildly impaired on a cognitive test or a clinical diagnosis of cognitive impairment ranging from mild cognitive impairment (MCI) or mild dementia (of any form). Mild dementia is the top end of this clinical diagnosis range. MCI is the low end of the range.
* reports <150 minutes of moderate to vigorous physical activity per week as per a single-item screener;
* self-reported ability to safely engage in regular walking;
* smartphone owner of a compatible smartphone for ≥1 month;
* willing and available second family member/friend/caregiver who owns a smartphone and can attend training sessions; and
* observed ability to reliably access and operate a smartphone during training.

Exclusion Criteria - Target User:

* unwillingness to meet at local community venues and/or via online meetings
* unwillingness to comply with study procedures for the length of the study
* inability to participate in English.
* residing outside of the local Los Angeles (LA) area and do not have the capacity to participate remotely or commuting to the University of Southern California (USC) study site
* recent cognitive status does not fall within an acceptable MCI/mild dementia range as determined through Montreal Cognitive Assessment (MoCA) if diagnosis was unverified by health care provider or by ADRC or memory and thinking problems were self-reported
* recent cognitive status is below what is acceptable for MCI/mild dementia as determined through MoCA if diagnosis was verified by health care provider or ADRC

Inclusion Criteria - Study Partner:

* English-speaking
* Family member/friend/caregiver of target user
* Owns a smartphone
* Willing to attend training sessions

Note: age limit criterion for target users does not apply to study partners

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-12-05 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 59 target users screened for eligibility; 15 signed consent; 15 completed the 2-month trial and included in analyses.
  6 study partners were screened for eligibility; 6 signed consent; 6 completed their role in the study. Only limited baseline analyses regarding characteristics were included.
Groups:
- Target Users - Moving Up-A App: In this single-arm trial, participants will use a physical activity smartphone app for a two-month period. The app includes motivational messages, tips to increase the intensity level of everyday activities, and strategies to reduce sedentary behaviors. Users can also track their physical activity levels and sedentary activity.
  Moving Up - A: Moving Up - A is a physical activity smartphone app for persons with mild cognitive impairment or mild forms of dementia. The app includes a personally tailored set of messages, tips, strategies, and tasks designed to increase physical activity levels and disrupt extended periods of sedentary time. Users also have the ability to track their steps and and sedentary behavior time as well as their progress towards activity goals.
- Study Partners - Moving Up-A App: Study partners: target users (participants) were invited to have a study partner (friend, family, caregiver) to support use of the Moving Up-A app by the target users.
Period: Overall Study
Arm/Group | Target Users - Moving Up-A App | Study Partners - Moving Up-A App
Started | 15 | 6
Completed | 15 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Target users' data were primarily collected and analyzed for this study. Only limited baseline data relevant to the study partners was collected and analyzed.
Groups:
- 2-month Pilot Test - Target Users: In this single-arm trial, participants will use a physical activity smartphone app for a two-month period. The app includes motivational messages, tips to increase the intensity level of everyday activities, and strategies to reduce sedentary behaviors. Users can also track their physical activity levels and sedentary activity.
  Moving Up - A: Moving Up - A is a physical activity smartphone app for persons with mild cognitive impairment or mild forms of dementia. The app includes a personally tailored set of messages, tips, strategies, and tasks designed to increase physical activity levels and disrupt extended periods of sedentary time. Users also have the ability to track their steps and and sedentary behavior time as well as their progress towards activity goals.
- 2-month Pilot Test - Study Partners: Target users (participants) were invited to have study partners to support use of the Moving Up-A app.
- Total: Total of all reporting groups
Arm/Group | 2-month Pilot Test - Target Users | 2-month Pilot Test - Study Partners | Total
Number analyzed (Participants) | 15 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only target user (not study partner) data were collected and analyzed for this baseline measure.
  years
    number analyzed (Participants) | 15 | 0 | 15
    (all) | 73.1 (4.7) |  | 73.1 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only target user (not study partner) data were collected and analyzed for this baseline measure.
  Participants
    number analyzed (Participants) | 15 | 0 | 15
    Hispanic or Latino | 0 |  | 0
    Not Hispanic or Latino | 15 |  | 15
    Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only target user (not study partner) data were collected and analyzed for this baseline measure.
  Participants
    number analyzed (Participants) | 15 | 0 | 15
    American Indian or Alaska Native | 0 |  | 0
    Asian | 3 |  | 3
    Native Hawaiian or Other Pacific Islander | 1 |  | 1
    Black or African American | 0 |  | 0
    White | 11 |  | 11
    More than one race | 0 |  | 0
    Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 6 | 21
Relationship to target user [Count of Participants; unit: Participants] — Population: This baseline measure is only relevant to study partners and not target users.
  Participants
    number analyzed (Participants) | 0 | 6 | 6
    Adult child |  | 1 | 1
    Spouse/partner |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Daily Steps Change From Baseline to Month 2
Description: Step counts (objective physical activity) were measured using the activPAL thigh-worn accelerometer during a 96-hour monitoring period.
  Change is computed as the activPAL-tracked mean daily steps at Month 2 minus that value at baseline
Time Frame: baseline and 2 months
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Target Users - Moving Up-A App
Number analyzed (Participants) | 15
steps per day | 604.1 (2560.4)
Statistical Analysis 1: Comparison: Target Users - Moving Up-A App; Test type: Superiority; p = 0.376, t-test, 2 sided; Mean Difference (Final Values) = 604.07, 95% CI 2-sided [-813.815 to 2021.95], Standard Deviation 2560.36

2. Secondary Outcome: Daily Sitting Time (activPAL) Change From Baseline to Month 2
Description: Objective sedentary activity time was measured using the activPAL thigh-worn accelerometer during a 96-hour monitoring period. Expressed as average minutes/day.
  Change is computed as the activPAL-tracked mean minutes/day of sitting time at Month 2 minus that value at baseline.
Time Frame: baseline and 2 months
Measure: Mean (Standard Deviation); unit: sitting minutes/day
Arm/Group | Target Users - Moving Up-A App
Number analyzed (Participants) | 15
sitting minutes/day | -35.0 (172.2)
Statistical Analysis 1: Comparison: Target Users - Moving Up-A App; Test type: Superiority; p = .444, t-test, 2 sided; Mean Difference (Final Values) = -35.019, 95% CI 2-sided [-130.36 to 60.324], Standard Deviation 172.168

3. Secondary Outcome: App Usability Measured Using the User Version of the Mobile Application Rating Scale (uMARS)
Description: The Mobile App Rating Scale User Version (uMARS) was used to measure user satisfaction with the app, particularly participant's ratings for app quality. The uMARS includes a usability feedback subindex which is comprised of the average of item responses for 4 subsections (engagement, functionality, aesthetics, information), to yield a total quality score. Ratings are on a scale of 1 (low perceived quality, min) to 5 (high perceived quality, max).
Time Frame: Month 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Target Users - Moving Up-A App
Number analyzed (Participants) | 15
score on a scale | 3.997 (.541)

4. Secondary Outcome: App Usage Behavior
Description: Usage behavior is defined as the percentage of days the app was opened at least once across the 2-month trial period
Time Frame: from baseline through Month 2 (daily)
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Target Users - Moving Up-A App
Number analyzed (Participants) | 15
percentage of days | 94.6 (10.4)

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Study Partners - Moving Up-A App: Target users (participants) were invited to have a study partner support them in using the Moving Up-A app. Study partners were not actively intervened on during this trial.
Arm/Group | Target Users - Moving Up-A App | Study Partners - Moving Up-A App
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6
Other Adverse Events (participants affected / at risk) | 1/15 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Target Users - Moving Up-A App (N=15) | Study Partners - Moving Up-A App (N=6)
Skin irritation from tape (Skin and subcutaneous tissue disorders) | 1 (1) | NA — Participant reported skin irritation from the Tegederm tape used to adhere the activity monitor to the thigh.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT04950998/Prot_SAP_000.pdf